CLINICAL TRIAL: NCT02490228
Title: Effectivity and Safety Study of Trans-artificial-urethral Resection of Female Urethral Caruncle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xuesong Li, Clinical Professor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAURFUC
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Urethral Caruncle
Keywords: female; minimally invasive surgery

ARMS (1):
- surgical group (Other): transurethral resection of urethral caruncle
  Interventions: Procedure: TAURFUC

INTERVENTIONS:
Procedure: TAURFUC — female patients with urethral caruncle will receive transurethral resection combine with extension tube.

SUMMARY:
To explore the minimally invasive and exhaustive treatment of female urethral canruncle by using trans-artificial-urethral resection of the canruncle. The investigators plant to recruit patients using this surgical method and study the effectivity of this method.

ELIGIBILITY:
Inclusion Criteria:

- patient with urethral caruncle

Exclusion Criteria:

- recurrence urethral caruncle

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Operative time | Up to 6 months
Length of hospital stay | Up to 6 months
Estimated blood loss | Up to 6 months
pathological type | Up to 6 months
Complication incidence rate | Up to 6 months

SECONDARY OUTCOMES:
recurrence-free survival | Up to 12 months